CLINICAL TRIAL: NCT03950739
Title: An Open-label, Clinical Study to Evaluate the Safety and Tolerability of Treprostinil Inhalation Powder (TreT) in Subjects With Pulmonary Arterial Hypertension Currently Using Tyvaso
Brief Title: Open-label, Clinical Study to Evaluate the Safety and Tolerability of TreT in Subjects With PAH Currently Using Tyvaso
Acronym: BREEZE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TIP-PH-101
Record Dates: First submitted 2019-05-09; First posted 2019-05-15 (Actual); Results first posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-08

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: prostacyclin
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Intervention Model Description: Single-sequence in which subjects on a stable regimen of Tyvaso switched to a corresponding dose of TreT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tyvaso to TreT (Experimental): Each subject received a corresponding dose of TreT for 3 weeks during the Treatment Phase based on the subject's current stable Tyvaso dose.
  Interventions: Drug: Treprostinil Inhalation Powder

INTERVENTIONS:
Drug: Treprostinil Inhalation Powder — Treprostinil inhalation powder single-use cartridges containing either 32 or 48 micrograms of treprostinil per cartridge (QID)
  Other Names: TreT

SUMMARY:
This was a Phase 1b safety and tolerability single-sequence study in which PAH subjects on a stable regimen of Tyvaso switched to a corresponding dose of TreT.

DETAILED DESCRIPTION:
United Therapeutics Corporation (UTC) developed a combination drug-device product comprised of a dry powder formulation of Treprostinil Inhalation Powder (TreT) and a small, portable, dry powder inhaler. In this Phase 1b safety and tolerability study, patients with PAH on a stable dose of Tyvaso (6 to 12 breaths 4 times daily [QID]) were evaluated after switching to a corresponding dose of TreT. Patients underwent PK assessments, safety assessments, a 6-Minute Walk Test (6MWT), and questionnaires for satisfaction/preference for inhaled devices and patient-reported PAH symptoms and impact. Following 3 weeks of treatment with TreT, patients were offered the opportunity to participate in the Optional Extension Phase until the drug/device became commercially available.

ELIGIBILITY:
Inclusion Criteria:

1. Subject voluntarily gave informed consent to participate in the study.
2. Subject was aged 18 years or older at the time of signing informed consent.
3. Women of childbearing potential were those who had experienced menarche and who had not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or were not postmenopausal (defined as amenorrhea for at least 12 consecutive months). WOCBP must have been nonpregnant (as confirmed by a urine pregnancy test at Screening prior to initiating study medication), nonlactating, and did 1 of the following:

   1. Abstained from intercourse (when it was in line with their preferred and usual lifestyle), or
   2. Used 2 medically acceptable, highly effective forms of contraception for the duration of study, and at least 30 days after discontinuing TreT. Medically acceptable, highly effective forms of contraception included approved hormonal contraceptives (oral, injectable, and implantable), intrauterine devices or systems, and barrier methods (such as a condom or diaphragm) when used with a spermicide.
4. Males with a partner of childbearing potential must have used a condom for the duration of treatment and for at least 48 hours after discontinuing TreT.
5. Subject was diagnosed with PAH as defined by the following World Health Organization (WHO) Group 1 categories:

   1. Idiopathic/familial
   2. Associated with unrepaired or repaired congenital systemic-to-pulmonary shunts (repaired ≥5 years prior to Screening)
   3. Associated with collagen vascular disease
   4. Associated with human immunodeficiency virus
   5. Associated with appetite suppressant/other drug or toxin use
6. Subject must have started Tyvaso ≥3 months prior to the Baseline Visit and was currently on a stable regimen (no change in dose within 30 days of Baseline Visit) of Tyvaso (6 to 12 breaths QID).
7. Baseline 6MWD ≥150 m.
8. If the subject was currently receiving other approved background therapy (eg, endothelin receptor antagonist or phosphodiesterase type 5 inhibitor or both), the subject must have been on a stable dose with no additions or discontinuations for a minimum of 30 days prior to Screening.
9. The subject had evidence of forced expiratory volume in 1 second (FEV1) ≥60% and FEV1/forced vital capacity ratio ≥60% during the 6 months prior to enrollment.
10. In the opinion of the Investigator, the subject was able to communicate effectively with study personnel, and was considered reliable, willing, and likely to be cooperative with protocol requirements, including all study visits.

Exclusion Criteria:

1. Subject was pregnant or lactating.
2. Subject was diagnosed with pulmonary hypertension for reasons other than WHO Group 1 as outlined in Inclusion Criterion 5 (including but not limited to portal hypertension, chronic thromboembolic disease, pulmonary veno-occlusive disease, hemolytic anemia, sarcoidosis).
3. Subject had a history of uncontrolled sleep apnea, parenchymal lung disease, or hemodynamically significant left-sided heart disease (including but not limited to aortic or mitral valve disease, pericardial constriction, restrictive or congestive cardiomyopathy, or coronary artery disease).
4. Subject was currently taking any other prostacyclin analogue or agonist, including but not limited to selexipag, epoprostenol, iloprost, or beraprost; except for acute vasoreactivity testing.
5. Subject experienced an acute exacerbation of disease or hospitalization for any reason within 30 days of the Screening Visit or between Screening and Baseline.
6. Subject was WHO Functional Class IV at Screening.
7. Subject had used any investigational drug/device or participated in any other investigational study with therapeutic intent within 30 days prior to the Screening Visit.
8. Subject had a history of anaphylaxis, a documented hypersensitivity reaction, or a clinically significant idiosyncratic reaction to treprostinil or excipients in the investigational product.
9. Subject had conditions that, in the opinion of the Investigator, would make the subject ineligible.
10. Subject was not able to perform inhalation maneuvers that met inspiratory training criteria.
11. Subject had a musculoskeletal disorder (eg, arthritis affecting the lower limbs, recent hip or knee joint replacement) or any disease that would likely be the primary limit to ambulation, or was connected to a machine that was not portable enough to allow for a 6MWT.
12. Subject had a new type of chronic therapy (including but not limited to oxygen, a different class of vasodilator, diuretic, and digoxin) for pulmonary hypertension added within 30 days of the Screening Phase.
13. Initiation of pulmonary rehabilitation within 12 weeks prior to the Baseline Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2023-08-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Department of Veterans Affairs Greater Los Angeles Healthcare System, Los Angeles, California
  - Ascension / St. Vincent's Lung Institute, Jacksonville, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of South Florida Center for Advanced Lung Disease, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Emory University Hospital, Atlanta, Georgia
  - The University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville Clinical Trials Unit, Louisville, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - University of Maryland Medical Center Division of Cardiology, Baltimore, Maryland
  - Penn Medicine University City, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Pulmonary Associates of Richmond, Inc., Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sahay S, Palevsky H, El-Kersh K, Restrepo-Jaramillo R, Bajwa AA, Desai S, Joly JM, Spikes LA, Eggert MS, Johri S, Shapiro SM, Fisher MR, Shah TG, Ramani GV, Mehta JP, Thrasher CM, Deng C, Smith P, Broderick M, Burger CD. BREEZE Optional Extension Phase: Long-term safety and efficacy of treprostinil dry powder inhaler (Tyvaso DPI) in pulmonary arterial hypertension. Respir Med. 2025 Nov;248:108318. doi: 10.1016/j.rmed.2025.108318. Epub 2025 Aug 27. PMID 40882760
- [Derived] Spikes LA, Bajwa AA, Burger CD, Desai SV, Eggert MS, El-Kersh KA, Fisher MR, Johri S, Joly JM, Mehta J, Palevsky HI, Ramani GV, Restrepo-Jaramillo R, Sahay S, Shah TG, Deng C, Miceli M, Smith P, Shapiro SM. BREEZE: Open-label clinical study to evaluate the safety and tolerability of treprostinil inhalation powder as Tyvaso DPI in patients with pulmonary arterial hypertension. Pulm Circ. 2022 Apr 7;12(2):e12063. doi: 10.1002/pul2.12063. eCollection 2022 Apr. PMID 35514770

RESULTS

PARTICIPANT FLOW:
Period: Treatment Phase
Arm/Group | Tyvaso to TreT
Started | 51
Completed | 49
Not Completed | 2
Not completed — Adverse Event | 2
Period: Optional Extension Phase
Arm/Group | Tyvaso to TreT
Started | 49
Completed | 31
Not Completed | 18
Not completed — Death | 1
Not completed — Progressive Disease | 5
Not completed — Adverse Event | 7
Not completed — Lost to Follow-up | 2
Not completed — Site Closure | 2
Not completed — Pregnancy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tyvaso to TreT
Number analyzed (Participants) | 51
Age, Continuous [Median (Full Range); unit: years] | 57.0 [23 to 82]
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 38
  ≥65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 47
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 51
Time Since PAH Diagnosis [Median (Full Range); unit: years] | 7.820 [0.49 to 30.88]
Current PAH Diagnosis [Count of Participants; unit: Participants]
  Idiopathic/Familial | 29
  Associated with Unrepaired or Repaired Congenital Systemic-to-Pulmonary Shunts | 4
  Associated with Collagen Vascular Disease | 14
  Associated with HIV | 1
  Associated with Appetite Suppressant/Other Drug or Toxin Use | 3
WHO Functional Class at Screening [Count of Participants; unit: Participants] — I: PH but without limitation of physical activity; physical activity without undue dyspnea or fatigue, chest pain or near syncope.
  II: PH with slight limitation of physical activity; physical activity causes undue dyspnea or fatigue, chest pain or near syncope.
  III: PH with marked limitation of physical activity; less than ordinary activity causes undue dyspnea or fatigue, chest pain or near syncope.
  IV: PH with inability to carry out any physical activity without symptoms. Signs of right heart failure. Dyspnea and/or fatigue at rest. Discomfort is increased by any physical activity.
  Participants
    I | 6
    II | 31
    III | 14
Background PAH Medications [Number; unit: participants]
  Endothelin receptor antagonist | 43
  Phosphodiesterase type 5 inhibitor | 41
  Soluble guanylate cyclase | 7
  No background PAH medication | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in 6-Minute Walk Distance (6MWD) From Baseline to Week 3
Description: 6MWD was evaluated at study entry and after 3 weeks of treatment with TreT.
Time Frame: From Baseline to 3 weeks of treatment with TreT
Population: Safety Population with 6MWD measurements at Week 3
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Tyvaso to TreT
Number analyzed (Participants) | 46
meters | 11.5 (32.9)

2. Primary Outcome: Subject Satisfaction With and Preference for Inhaled Treprostinil Devices
Description: Subject satisfaction with and preference for the inhaled treprostinil device was evaluated with the Preference Questionnaire for Inhaled Treprostinil Devices (PQ-ITD). The PQ-ITD is a questionnaire given to evaluate subject satisfaction with and preference for inhaled treprostinil devices. The questionnaire provides 12 different statements around inhaled device satisfaction and allows for 5 response options: strongly disagree, disagree, neutral, agree, and strongly agree.
Time Frame: After 3 weeks of treatment with TreT (after switching from the Tyvaso Inhalation System)
Population: Safety Population with PQ-ITD responses at Week 3
Measure: Count of Participants; unit: Participants
Arm/Group | Tyvaso to TreT
Number analyzed (Participants) | 46
Participants
  Strongly Disagree | 0
  Disagree | 0
  Neutral | 1
  Agree | 5
  Strongly Agree | 40

3. Primary Outcome: Change in Patient-reported PAH Symptoms and Impact From Baseline to Week 3
Description: Patient-reported PAH symptoms and impact were evaluated with the PAH Symptoms and Impact (PAH-SYMPACT) Questionnaire. The PAH-SYMPACT is a 23-item patient-reported outcome questionnaire that consists of 11 symptom items, 11 impact items, and 1 item on oxygen use. The symptom items are divided into cardiopulmonary and cardiovascular domains, and the impact items are divided into physical and emotional/cognitive domains. Symptom and impact domain scores (range 0 to 4) are calculated as the sum of the scores for the items included in the domain divided by the number of items in the domain.
  For all domains, a higher score indicates more severe symptoms/impacts.
Time Frame: From Baseline to 3 weeks of treatment with TreT
Population: Safety Population with PAH-SYMPACT scores at Week 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tyvaso to TreT
Number analyzed (Participants) | 46
score on a scale
  Cardiopulmonary Symptoms Domain Score | -0.05 (0.27)
  Cardiovascular Symptoms Domain Score | -0.06 (0.33)
  Physical Impacts Domain Score | -0.14 (0.46)
  Cognitive/Emotional Impacts Domain Score | -0.17 (0.40)

4. Primary Outcome: Change in Patient-reported PAH Symptoms and Impact From Baseline to Week 11 (for Subjects Participating in the OEP)
Description: as for outcome 3
Time Frame: From Baseline to 11 weeks of treatment with TreT
Population: Safety Population with PAH-SYMPACT scores at Week 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tyvaso to TreT
Number analyzed (Participants) | 37
score on a scale
  Cardiopulmonary Symptoms Domain Score | -0.04 (0.36)
  Cardiovascular Symptoms Domain Score | -0.05 (0.40)
  Physical Impacts Domain Score: number analyzed (Participants) | 36
  Physical Impacts Domain Score | -0.20 (0.59)
  Cognitive/Emotional Impacts Domain Score: number analyzed (Participants) | 36
  Cognitive/Emotional Impacts Domain Score | -0.13 (0.51)

ADVERSE EVENTS:
Time Frame: All AEs were documented from the time of informed consent until the time screen failure was documented, until the subject either discontinued from the study, or the End of Study (EOS)/Early Termination (ET) assessments were completed, up to 201.1 weeks.
Description: All AEs were followed until either resolution (or return to normal or baseline values), until they were judged by the Investigator to no longer be clinically significant, the subject was lost to further follow-up, or for at least 30 days if the AE extended beyond the EOS/ET Visit. All SAEs that occurred during the study were followed until resolution, death, or the subject was lost to follow-up, even if they were ongoing more than 30 days after completion of the final study visit.
Groups:
- Tyvaso to TreT 32 mcg (Treatment Phase); Tyvaso to TreT 48 mcg (Treatment Phase); Tyvaso to TreT 64 mcg (Treatment Phase); Tyvaso to TreT 32 mcg (Optional Extension Phase); Tyvaso to TreT 48 mcg (Optional Extension Phase); Tyvaso to TreT 64 mcg (Optional Extension Phase): Each subject received a corresponding dose of TreT for 3 weeks during the Treatment Phase based on the subject's current stable Tyvaso dose.
  Treprostinil Inhalation Powder: Treprostinil inhalation powder single-use cartridges containing either 32 or 48 micrograms of treprostinil per cartridge (QID)
Arm/Group | Tyvaso to TreT 32 mcg (Treatment Phase) | Tyvaso to TreT 48 mcg (Treatment Phase) | Tyvaso to TreT 64 mcg (Treatment Phase) | Tyvaso to TreT 32 mcg (Optional Extension Phase) | Tyvaso to TreT 48 mcg (Optional Extension Phase) | Tyvaso to TreT 64 mcg (Optional Extension Phase)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/27 | 0/22 | 0/2 | 0/26 | 1/21
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/27 | 1/22 | 1/2 | 12/26 | 12/21
Other Adverse Events (participants affected / at risk) | 0/2 | 17/27 | 14/22 | 2/2 | 25/26 | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tyvaso to TreT 32 mcg (Treatment Phase) (N=2) | Tyvaso to TreT 48 mcg (Treatment Phase) (N=27) | Tyvaso to TreT 64 mcg (Treatment Phase) (N=22) | Tyvaso to TreT 32 mcg (Optional Extension Phase) (N=2) | Tyvaso to TreT 48 mcg (Optional Extension Phase) (N=26) | Tyvaso to TreT 64 mcg (Optional Extension Phase) (N=21)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Parotitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rocky mountain spotted fever (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ureteric injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oestrogen receptor assay positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adult failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug dependence (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Renal mass (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tyvaso to TreT 32 mcg (Treatment Phase) (N=2) | Tyvaso to TreT 48 mcg (Treatment Phase) (N=27) | Tyvaso to TreT 64 mcg (Treatment Phase) (N=22) | Tyvaso to TreT 32 mcg (Optional Extension Phase) (N=2) | Tyvaso to TreT 48 mcg (Optional Extension Phase) (N=26) | Tyvaso to TreT 64 mcg (Optional Extension Phase) (N=21)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 11 (11) | 7 (7) | 1 (2) | 4 (4) | 4 (5)
Headache (Nervous system disorders) | 0 (0) | 4 (4) | 4 (4) | 2 (3) | 6 (8) | 4 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 10 (12) | 4 (4)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 4 (6)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 4 (5) | 4 (6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 1 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 5 (9)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (4)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (3) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 3 (3)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (5)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 3 (3)
Myaligia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 6 (6) | 2 (3)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 1 (2)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and/or Principal Investigator agree not to publish or publicly present any results of the Study without the prior written consent of Sponsor, not to be unreasonably withheld or delayed. Institution and/or Principal Investigator further agree to provide Sponsor with drafts of any such publication or presentation for review and approval no less than 30 days prior to submission for publication or the date of public presentation.

DOCUMENTS (2):
  • Study Protocol (2020-04-02): https://cdn.clinicaltrials.gov/large-docs/39/NCT03950739/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/39/NCT03950739/SAP_001.pdf